CLINICAL TRIAL: NCT06338891
Title: Can Gluten/Wheat or Other Foods be Responsible for FMF Attacks: A Survey on Self-perceived Food Sensitivity in FMF Patients
Brief Title: Can Gluten/Wheat or Other Foods be Responsible for FMF Attacks
Status: Recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Associate Professor, University of Palermo
Other Study IDs: ACPM34
Record Dates: First submitted 2024-02-26; First posted 2024-04-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Familial Mediterranean Fever; Non-celiac Gluten Sensitivity
Keywords: Familial Mediterranean Fever; Non-celiac Gluten Sensitivity
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FMF patients: Patients, of both sexes, aged between 6 months and 80 years, affected by FMF, classified according to the Eurofever/PRINTO criteria
  Interventions: Other: Main questionnaire; Other: Secondary questionnaire
- Control subjects: Subjects of the vaccination center of the University Hospital 'Paolo Giaccone'" of Palermo, Italy
  Interventions: Other: Secondary questionnaire

INTERVENTIONS:
Other: Main questionnaire — Main questionnaire will evaluate the demographic and genetic characteristics, clinical manifestations, and self-perception of sensitivity to wheat or other food and the possible relationship between the intake of wheat or other foods and the flare-ups of the disease in FMF patients
  Groups: FMF patients
Other: Secondary questionnaire — Secondary questionnaire will investigate the possible appearance of gastrointestinal and extraintestinal symptoms linked to the ingestion of gluten/wheat, which are not identifiable, by the patient, as FMF flare-ups, but might be compatible with a NCGS/NCWS diagnosis

SUMMARY:
Familial Mediterranean Fever (FMF) is a chronic hereditary autoinflammatory disease caused by mutations in the MEditerranean FeVer (MEFV) gene which codes for pyrin. Dysfunction of this protein determines an inappropriate response to inflammatory stimuli. The clinical course of the disease is characterized by recurrent episodes of fever and inflammation of the serous membranes, which manifest with chest, abdominal and joint pain. Several studies suggest a possible association between acute FMF attacks and dietary triggers, including wheat. However, it is still unclear to what extent wheat is responsible for the reactivation of FMF and if, between one acute attack and another, patients with FMF experience other symptoms, both gastrointestinal and extraintestinal, characteristic of gluten/wheat sensitivity not linked to celiac disease or immunoglobulin E (IgE)-mediated wheat allergy (i.e. Non-Celiac Wheat Gluten/Sensitivity, NCGS/NCWS).

Therefore, this study aims to evaluate the appearance of symptoms compatible with an acute attack of FMF following the ingestion of wheat or other foods, and the prevalence of self-perceived gluten/wheat sensitivity in patients with FMF.

DETAILED DESCRIPTION:
Familial Mediterranean Fever (FMF) is a hereditary autoinflammatory disease, with autosomal recessive transmission, secondary to the mutation of the MEFV (MEditerranean FeVer) gene. Several mutations have been identified as responsible for the dysfunction of pyrin, a protein involved in the regulation of inflammatory processes. The resulting inappropriate inflammatory response generally manifests with recurrent and short-lasting episodes of fever, associated with inflammation of the serosa (FMF "attack"). Among the most commonly reported symptoms during an acute attack, abdominal pain prevails, which is often the first symptom to appear. The most fearful complication of this pathology is amyloidosis. Currently, the first-line treatment for symptom control and prevention of amyloidosis is colchicine. However, despite treatment, FMF attack may still occur following exposure to some triggers, such as, for example, infections, trauma, physical activity, and stress. Various researchers have also evaluated dietary habits and the intake of certain foods, such as, for example, a diet rich in fats, cow's milk, and wheat, as possible triggers of the FMF attacks.

Little is known about the trigger effect of foods on the exacerbation of FMF and the evidence from the few studies in the literature appears to be controversial. The results relating to the protective effect of a low-fat and a low-salt diet on the exacerbation of symptoms in patients with FMF are conflicting. Furthermore, in a prospective study, conducted on a limited sample of patients with FMF, it was demonstrated that the ingestion of wheat could be responsible for both the clinical (with worsening of the disease activity score), and the immunological reactivation of the disease [with evidence of increased levels of serum C-reactive protein (CRP), serum amyloid A (SSA), and circulating cluster of differentiation (CD)14+/IL1Beta+ and CD14+/TNFalpha+ monocytes]. The macronutrients in wheat potentially responsible for activating the immune system could be gluten and/or alpha-amylase/trypsin inhibitors Amylase-Trypsin Inhibitors (ATIs). Some researchers hypothesize that these protein components of wheat are also responsible for an alteration of the intestinal microbiota, which, in turn, by alteration of intestinal permeability and translocation of bacterial products, can lead to the activation of the immune system, both innate and adaptive, at a local and a systemic level, and, therefore, to the worsening of the inflammatory state of patients with autoinflammatory/autoimmune diseases. Indeed, in patients with FMF, several studies evaluated the relationship between modifications in intestinal microbiota and disease activity. For example, one study demonstrated the presence of mucosal damage predominantly affecting the jejunum and terminal ileum in approximately half of a group of 41 patients with FMF undergoing endoscopic examinations. This finding would determine the translocation and dissemination of molecules associated with pathogens and mucosal damage (Pathogen Associated Molecular Patterns (PAMPs), and , Damage Associated Molecular Patterns (DAMPs)) capable of triggering the acute attacks of the disease. Furthermore, it has been shown that the overgrowth of intestinal bacterial flora (better known as Small Intestinal Bacterial Overgrowth (SIBO), causing the blood diffusion of bacterial metabolism products, can alter the response to colchicine and cause poor control of disease activity, thus suggesting that the gut microbiota can modulate both the clinical expression and the therapeutic response of FMF. In turn, in these patients, alterations of microbiota and, consequently, of intestinal permeability, could depend both on the chronic inflammatory state of the disease itself and on extrinsic factors (i.e. dietary ones).

To date there are only few data regarding the relationship between ingestion of wheat and other foods and the flare-ups of the FMF and the prevalence of gluten/wheat sensitivity not linked to celiac disease or IgE-mediated allergy to wheat Non-Celiac Gluten/Wheat Sensitivity (NCGS/NCWS) in patients with FMF. Therefore, the aims of this study are:

1. To evaluate, in patients with a definite diagnosis of FMF, the prevalence of the trigger effect of wheat or other foods other than wheat, defined as the appearance of symptoms and signs, identifiable as reactivation of FMF, after ingestion of wheat or other specific foods.
2. To identify possible demographic, clinical and genetic differences between FMF patients without and with reported trigger effects of wheat or other specific foods.
3. To evaluate, in patients with a definite diagnosis of FMF, the prevalence of self-perception NCGS/NCWS, defined as the appearance of gastrointestinal and extraintestinal symptoms caused by the ingestion of gluten/wheat, compared to a control group [subjects of the vaccination center of the University Hospital 'Paolo Giaccone'" of Palermo, Italy].
4. To identify demographic, clinical, and genetic differences between FMF patients without and with self-reported NCGS/NCWS.

ELIGIBILITY:
Inclusion Criteria:

* Patients, of both sexes, aged between 6 months and 80 years, affected by FMF, classified according to the Eurofever/PRINTO criteria.
* Patients able to understand and complete the questionnaires independently (or, in the case of pediatric ones, analyzed through the answers provided by parents).

Exclusion Criteria:

* Patients aged <6 months and >80 years.
* Patients unable to provide informed consent or complete the questionnaires.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of FMF will be enrolled in four Italian centers: the "Ambulatorio di Celiachia ed Intolleranze Alimentari" of "Azienda Ospedaliera Universitaria Policlinico (AOUP) 'Paolo Giaccone'", Palermo, Italy, the Internal Medicine Unit of "Azienda Ospedaliera 'Ospedali Riuniti Villa Sofia-Cervello'", Palermo, Italy, the "Centro di Riferimento per le Malattie Autoinfiammatorie e per le Malattie Lisosomiali" and the "Unità Malattie Rare, Centro Ricerca sulle Febbri Periodiche" of "Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS", Rome, Italy. Patients will be asked to reposnd to a main questionnaire, to evaluate the patient's demographic, clinical and genetic characteristics, and the perception of a link between FMF exacerbations and intake of wheat or other foods, and, in patients with self-reported NCGS/NCWS, gastrointestinal and extraintestinal manifestations related to gluten/wheat intake will be investigated using a further secondary questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the self-perception of wheat as a potential trigger of acute attack in patients with familial Mediterranean fever (FMF) | From May 2024 to May 2025
  To determine the prevalence of the self-perception of wheat as a potential trigger of acute attack in patients with FMF, defined as the appearance of symptoms and signs compatible with FMF flare-up following wheat intake.
Prevalence of the self-perception of other foods, other than wheat, as potential triggers of an acute attack in patients with FMF | From May 2024 to May 2025
  To determine the prevalence of the self-perception of other foods, other than wheat, as potential triggers of an acute attack in patients with FMF, defined as the appearance of symptoms and signs compatible with a flare-up of FMF following the intake of these specific foods, other than wheat.
Prevalence of self-reported NCGS/NCWS in patients with FMF | From May 2024 to May 2025
  To determine the prevalence of self-reported NCGS/NCWS in patients with FMF, defined as the appearance of gastrointestinal and extraintestinal symptoms and signs secondary to gluten/wheat ingestion, compatible with the clinical manifestations of NCGS/NCWS and not identifiable, by the patient, as FMF flare-ups, compared to a control group.

SECONDARY OUTCOMES:
Genetic differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in prevalence in the specific genetic mutations related to FMF between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Genetic differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in prevalence in the specific genetic mutations related to FMF between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Genetic differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in prevalence in the specific genetic mutations related to FMF between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Ethnic group differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in ethnic group prevalence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Ethnic group differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in ethnic group prevalence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Ethnic group differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in ethnic group prevalence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Education level differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in education level prevalence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Education level differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in education level prevalence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Education level differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in education level prevalence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Working activity differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in working activity between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Working activity differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in working activity between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Working activity differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in working activity between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Gastrointestinal symptoms differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms prevalence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Gastrointestinal symptoms differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms prevalence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Gastrointestinal symptoms differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms prevalence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Extraintestinal symptoms differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms prevalence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Extraintestinal symptoms differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms prevalence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Extraintestinal symptoms differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms prevalence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Extraintestinal symptoms duration differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms duration between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Extraintestinal symptoms duration differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms duration between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Extraintestinal symptoms duration between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in extraintestinal symptoms duration between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Gastrointestinal symptoms duration differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms duration between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Gastrointestinal symptoms duration differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms duration between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Gastrointestinal symptoms duration differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in gastrointestinal symptoms duration between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
FMF specific drugs intake differences between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
FMF specific drugs intake differences between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
FMF specific drugs intake differences between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Differences in number/year of FMF attacks between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in number/year of FMF attacks between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in number/year of FMF attacks between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in number/year of FMF attacks between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in number/year of FMF attacks between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in number/year of FMF attacks between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Differences in FMF specific drugs intake adherence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake adherence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in FMF specific drugs intake adherence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake adherence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in FMF specific drugs intake adherence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in FMF specific drugs intake adherence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Differences in marital status between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in marital status prevalence between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in marital status between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in marital status prevalence between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in marital status between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in marital status prevalence between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Differences in age at FMF diagnosis between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in age at FMF diagnosis between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in age at FMF diagnosis between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in age at FMF diagnosis between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in age at FMF diagnosis between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in age at FMF diagnosis between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.
Differences in age at FMF symptom's onset between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. | From May 2024 to May 2025
  To define any difference in age at FMF symptom's onset between FMF patients who perceive a trigger effect of wheat and those who do not identify this specific food as a potential trigger of the disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in age at FMF symptom's onset between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. | From May 2024 to May 2025
  To define any difference in age at FMF symptom's onset between FMF patients who perceive a trigger effect of foods other than wheat and those who do not identify foods other than wheat as a potential trigger of disease flares. The data will be collected through the answers provided to the questions in the main questionnaire.
Differences in age at FMF symptom's onset between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. | From May 2024 to May 2025
  To define any difference in age at FMF symptom's onset between patients with FMF who self-report NCGS/NCWS and those who do not self-report it. The data will be collected through the answers provided to the questions in the secondary questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Director — University of Palermo
Locations (1):
- University Hospital of Palermo, Palermo, Sicily, Italy

REFERENCES:
- [Background] Carroccio A, Mansueto P, Soresi M, Fayer F, Di Liberto D, Monguzzi E, Lo Pizzo M, La Blasca F, Geraci G, Pecoraro A, Dieli F, Schuppan D. Wheat Consumption Leads to Immune Activation and Symptom Worsening in Patients with Familial Mediterranean Fever: A Pilot Randomized Trial. Nutrients. 2020 Apr 17;12(4):1127. doi: 10.3390/nu12041127. PMID 32316660
- [Background] Demir A, Akyuz F, Gokturk S, Evirgen S, Akyuz U, Ormeci A, Soyer O, Karaca C, Demir K, Gundogdu G, Gulluoglu M, Erer B, Kamali S, Kaymakoglu S, Besisik F, Gul A. Small bowel mucosal damage in familial Mediterranean fever: results of capsule endoscopy screening. Scand J Gastroenterol. 2014 Dec;49(12):1414-8. doi: 10.3109/00365521.2014.976838. Epub 2014 Nov 5. PMID 25369738
- [Background] Deshayes S, Fellahi S, Bastard JP, Launay JM, Callebert J, Fraisse T, Buob D, Boffa JJ, Giurgea I, Dupont C, Jegou S, Straube M, Karras A, Aouba A, Grateau G, Sokol H, Georgin-Lavialle S; AA Amyloidosis Study Group; AA amyloidosis Study Group. Specific changes in faecal microbiota are associated with familial Mediterranean fever. Ann Rheum Dis. 2019 Oct;78(10):1398-1404. doi: 10.1136/annrheumdis-2019-215258. Epub 2019 Aug 3. PMID 31377728
- [Background] Ekinci RMK, Balci S, Bisgin A, Cetin FT, Tumgor G. The contribution of diet preference to the disease course in children with familial Mediterranean fever: a cross-sectional study. Reumatologia. 2020;58(2):81-86. doi: 10.5114/reum.2020.95361. Epub 2020 Apr 30. PMID 32476680
- [Background] Gattorno M, Hofer M, Federici S, Vanoni F, Bovis F, Aksentijevich I, Anton J, Arostegui JI, Barron K, Ben-Cherit E, Brogan PA, Cantarini L, Ceccherini I, De Benedetti F, Dedeoglu F, Demirkaya E, Frenkel J, Goldbach-Mansky R, Gul A, Hentgen V, Hoffman H, Kallinich T, Kone-Paut I, Kuemmerle-Deschner J, Lachmann HJ, Laxer RM, Livneh A, Obici L, Ozen S, Rowczenio D, Russo R, Shinar Y, Simon A, Toplak N, Touitou I, Uziel Y, van Gijn M, Foell D, Garassino C, Kastner D, Martini A, Sormani MP, Ruperto N; Eurofever Registry and the Paediatric Rheumatology International Trials Organisation (PRINTO). Classification criteria for autoinflammatory recurrent fevers. Ann Rheum Dis. 2019 Aug;78(8):1025-1032. doi: 10.1136/annrheumdis-2019-215048. Epub 2019 Apr 24. PMID 31018962
- [Background] Leccioli V, Oliveri M, Romeo M, Berretta M, Rossi P. A New Proposal for the Pathogenic Mechanism of Non-Coeliac/Non-Allergic Gluten/Wheat Sensitivity: Piecing Together the Puzzle of Recent Scientific Evidence. Nutrients. 2017 Nov 2;9(11):1203. doi: 10.3390/nu9111203. PMID 29099090
- [Background] Mansueto P, Seidita A, Chiavetta M, Genovese D, Giuliano A, Priano W, Carroccio A, Casuccio A, Amodio E. Familial Mediterranean Fever and Diet: A Narrative Review of the Scientific Literature. Nutrients. 2022 Aug 5;14(15):3216. doi: 10.3390/nu14153216. PMID 35956392
- [Background] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Background] MELLINKOFF SM, SCHWABE AD, LAWRENCE JS. A dietary treatment for familial Mediterranean fever. Arch Intern Med. 1961 Jul;108:80-5. doi: 10.1001/archinte.1961.03620070082010. No abstract available. PMID 13769243
- [Background] Schwabe AD, Peters RS. Familial Mediterranean Fever in Armenians. Analysis of 100 cases. Medicine (Baltimore). 1974 Nov;53(6):453-62. doi: 10.1097/00005792-197411000-00005. No abstract available. PMID 4437392
- [Background] Uhde M, Ajamian M, Caio G, De Giorgio R, Indart A, Green PH, Verna EC, Volta U, Alaedini A. Intestinal cell damage and systemic immune activation in individuals reporting sensitivity to wheat in the absence of coeliac disease. Gut. 2016 Dec;65(12):1930-1937. doi: 10.1136/gutjnl-2016-311964. Epub 2016 Jul 25. PMID 27459152
- [Background] Verrecchia E, Sicignano LL, La Regina M, Nucera G, Patisso I, Cerrito L, Montalto M, Gasbarrini A, Manna R. Small Intestinal Bacterial Overgrowth Affects the Responsiveness to Colchicine in Familial Mediterranean Fever. Mediators Inflamm. 2017;2017:7461426. doi: 10.1155/2017/7461426. Epub 2017 Dec 12. PMID 29379228
- [Background] Yenokyan G, Armenian HK. Triggers for attacks in familial Mediterranean fever: application of the case-crossover design. Am J Epidemiol. 2012 May 15;175(10):1054-61. doi: 10.1093/aje/kwr460. Epub 2012 Jan 10. PMID 22234484